CLINICAL TRIAL: NCT05556577
Title: Weight Cycle Impacted by Health Lifestyle Post Pharmacotherapy Intervention
Brief Title: Weight Cycle Post Intervention
Status: Withdrawn | Type: Observational
Why Stopped: duplicated registration
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-084
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: investigational medicine product (IMP) — Investigational medicine product (IMP) received at SURMOUNT-CN trial
Other: placebo — Placebo received at SURMOUNT-CN trial

SUMMARY:
The aim of this follow-up (FU) study is to examine trajectory of body weight impacted by self-reported diet patterns and physical activities in 6 months at 3 monthly intervals from treatment cessation among patients who completed a pharmacotherapy trial. In addition, patient self-reported diet patterns and physical activities at respective time points will be described.

DETAILED DESCRIPTION:
This is a real-world prospective observational study with primary data collection. All participants with a background be recommended to adopt lifestyle intervention as chronic weight management in China clinical practice. This FU study will enroll patients who completed SURMOUNT-CN trials, with planed study duration of 6 months. No investigational medicine is applied in this prospective follow-up study.

Patients are requested to report body weight, waist circumferences, blood pressure, diet, physical activities, and laboratory results if available, at 3 monthly intervals during the 6-month follow-up period. Patients are also asked if they receive any Anti-Obesity medication (AOM) or participate in any interventional clinical trials indicated for weight management during study period. Summary statistics will be respectively applied to examine changes from trial baseline (time at trial randomization, week 0) and study baseline (time at 52 weeks from trial randomization, week 52) to each scheduled follow-up (at week 65 and week 78) by study arms in SURMOUNT-CN trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients who completed SURMOUNT-CN trial are target patients. Those who consent to this follow-up study are study participants.

Exclusion Criteria:

* Those in the SURMOUNT-CN trial who denied to participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who completed SURMOUNT-CN trial are target patients. Those who consent to this follow-up study are study participants.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
the change in body weight | at week 65 and week 78 from study baseline

IPD SHARING:
Plan to Share IPD: No